CLINICAL TRIAL: NCT06404177
Title: Dexketoprofen ® IV Versus Piroxicam® IM in Emergency Pain Management
Brief Title: Enantyum® IV Versus Piroxen® IM in Emergency Pain Management
Acronym: PiDex
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Riadh Boukef (Other)
Responsible Party: Sponsor-Investigator, Riadh Boukef, professor, Hôpital Universitaire Sahloul
Organization: Hôpital Universitaire Sahloul (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexketoprofene-Piroxicam
Record Dates: First submitted 2023-07-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — dexketoprofen trometamol; Piroxicam

STUDY DESIGN:
Intervention Model Description: prospective, randomised , double blind controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexketoprofen (Experimental): Patients receive a perfusion of Dexketoprofen in intraveinous with an injection of istonic saline IM injection
  Interventions: Drug: Dexketoprofen
- Piroxicam (Active Comparator): Patients receive an intramuscular injection of piroxicam with an intravenous isotonic saline
  Interventions: Drug: Piroxicam

INTERVENTIONS:
Drug: Dexketoprofen — An intravenous perfusion of eunantyum with an intramuscular isotonic saline
  Other Names: Placebo IM
  Arms: Dexketoprofen
Drug: Piroxicam — intramuscular injection of piroxicam with a perfusion of isotonic saline intravenous
  Other Names: placebo IV
  Arms: Piroxicam

SUMMARY:
For pain of traumatic origin, the RICE protocol (Rest, Ice, Compression, Elevation) is the main therapeutic measure during the first 4 to 5 days post-trauma. However, there is currently insufficient evidence that this protocol is effective [4].

In the emergency department, paracetamol, NSAIDs or a combination of several molecules are generally prescribed. Patients even use these drugs without a prescription.

The aim of this study is to Compare the effect of dexketoprofen® IV versus piroxen® IM in the treatment of pain in emergency departments.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind, controlled study conducted at the Sahloul emergency department, Sousse.

Study duration: 3 months.

Inclusion criteria:

Patients over 18 years of age requiring analgesia for acute pain of traumatic origin and who signed a written consent form were included in this study.

Exclusion criteria:

Patients who meet the following conditions:

* refusal, incapacity, difficulties with consent or communication
* Patients with chronic pain.
* Any known allergy or secondary reaction to piroxen or dexketoprofen trometamol.
* Pregnant women.
* Cirrhosis of the liver.

Methodology:

1. Dexketoprofen group Patient receives an intravenous injection of Dexketoprofen + IM placebo + follow-up sheet + appointment card.
2. Piroxican group. Patients receive one intramuscular Piroxen injection + IV SSI infusion + follow-up sheet + appointment card.

For each patient included, VAS, blood pressure, heart rate, respiratory rate and Sa02 are taken on admission and discharge from the emergency department, and at the second telephone visit after 07 days.

At the 7th day visit (by telephone), patients were asked to answer satisfaction questions and complete the EQ50 quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who required analgesia for acute pain of traumatic origin and who signed a written consent form were included in the study.

Exclusion Criteria:

* Patients who meet the following conditions:
* refusal, incapacity, difficulties with consent or communication
* Patients with chronic pain.
* Any known allergy or secondary reaction to piroxen or dexketoprofen trometamol.
* Pregnant women.
* Cirrhosis of the liver.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to pain resolution | 120 minutes
  VAS<3

SECONDARY OUTCOMES:
rescue tratment | 120 minutes
  rate of the use of another analgesics
Side effects | 7 days
  number of patients with epigastralgia , digestive bleeding, nausea, vomiting
patient satisfaction | 7 days
  rate of satisfaction with likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sahloul University Hospital, Sousse, Tunisia